CLINICAL TRIAL: NCT03082339
Title: Influence of Cortisone on QTc-interval
Brief Title: Cortisone and QTc-Interval
Status: Completed | Type: Observational
Sponsor: Asklepios Neurological Clinic Bad Salzhausen (Other)
Collaborators: University of Giessen (Other)
Responsible Party: Sponsor
Other Study IDs: QTc25416
Record Dates: First submitted 2017-03-12; First posted 2017-03-17 (Actual); Last update posted 2020-05-04 (Actual); Status verified 2020-05

CONDITIONS: QTc-interval
MeSH Terms: interventions — Cortisone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Neurology: Patients with inflammatory disease, especially multiple sclerosis, who underwent therapy with cortisone (>=40mg/d)
  Interventions: Other: Cortisone
- Pulmonology: Patients after LTX (under medication possible prologing QTc-interval), who underwent therapy with cortisone (>=40mg/d)
  Interventions: Other: Cortisone

INTERVENTIONS:
Other: Cortisone — Observation of QTc-interval

SUMMARY:
Scientific and clinical data report about shortening of QTc-interval in patients treated with cortisone. Peal et al. analyzed chemical suppression of long QT syndrome (Type 2) in an in vivo zebrafish model. Their study revealed that flurandrenolide reproducibly suppressed the long QT phenotype via the glucocorticoid signaling pathway. In contrast to treatment with dexamethasone and testosterone, treatment with pure mineralocorticoid deoxycorticosterone acetate did not suppress long QT phenotype. Knockdown of the glucocorticoid receptor or, conversely, of the androgen receptor showed that flurandrenolide acting through the glucocorticoid receptor shortens ventricular action potentials. The mechanism is distinct from trafficking rescue of the defective zebrafish-ERG channel. The authors discuss that a drug normalizing repolarization would be a novel therapeutic tool in long QT syndrome and conclude that glucocorticoids could be expected to aid in the acute management of patients with long QT syndrome, e.g. in episodes of arrhythmic storm. In addition, corticoid induced normalization of the QT interval is reported in a patient with drug-induced prolongation of the QTc interval. Brostoff et al. report on a patient suffering from mucocutaneous leishmaniasis treated with sodium stibogluconate. During therapy, the QTc interval prolonged and returned to normal within 4 days after starting glucocorticoid therapy with prednisolone 20 mg twice daily.

Interrogation of the study:

* shortens cortisone the QTc-interval?
* how long is the interval until shortening of QTc-interval?
* is the effect prolonged?
* is the effect dose dependend?

ELIGIBILITY:
Inclusion Criteria:

* patients who underwent therapy with cortisone (>=40mg/d)

Exclusion Criteria:

* patients with elevated intracranial pressure
* myocardial infarction within the last 6 months
* untreated stenosis of the coronary arteries
* right bundle branch block
* autoimmune disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with inflammatory neurological (especially multiple sclerosis) and pulmological (after LTX) diseases, who underwent therapy with cortisone (>= 40 mg/d).
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2020-04-25 (Actual); Study Completion 2020-04-25 (Actual)

PRIMARY OUTCOMES:
Duration of QTc-interval | 1 week
  daily ECG controls and measuring QTc-interval

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - University Giessen, Giessen
  - Neurologische Klinik Bad Salzhausen, Nidda

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Brostoff JM, Lockwood DN. Glucocorticoids as a novel approach to the treatment of disabling side effects of sodium stibogluconate. J Clin Pharm Ther. 2012 Feb;37(1):122-3. doi: 10.1111/j.1365-2710.2011.01259.x. Epub 2011 Apr 4. PMID 21457289
- [Background] Peal DS, Mills RW, Lynch SN, Mosley JM, Lim E, Ellinor PT, January CT, Peterson RT, Milan DJ. Novel chemical suppressors of long QT syndrome identified by an in vivo functional screen. Circulation. 2011 Jan 4;123(1):23-30. doi: 10.1161/CIRCULATIONAHA.110.003731. Epub 2010 Nov 15. PMID 21098441